CLINICAL TRIAL: NCT03252938
Title: An Explorative, Open-labeled, Phase I Study to Evaluate the Feasibility and the Safety of IMP321 in Combination With Immunotherapeutic/Targeted/Chemotherapeutic Agents or Via New Routes of Application in Advanced Stage Solid Tumors
Brief Title: Feasibility and Safety of IMP321 (Eftilagimod Alpha) for Advanced Stage Solid Tumors
Acronym: INSIGHT
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Institut für Klinische Krebsforschung IKF GmbH at Krankenhaus Nordwest (Other)
Collaborators: Immutep S.A.S. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INSIGHT
Record Dates: First submitted 2017-08-14; First posted 2017-08-17 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Solid Tumors; Peritoneal Carcinomatosis; NSCLC Adenocarcinoma; Urothelial Carcinoma
Keywords: solid tumor; peritoneal carcinomatosis
MeSH Terms: conditions — Peritoneal Neoplasms; Carcinoma, Transitional Cell | interventions — soluble LAG-3 protein, human; avelumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Solid tumors (Experimental): Biweekly intra-tumoral injections of escalating doses (6 mg, 12 mg, 24 mg and 30 mg) of IMP321 as a monotherapy (intratumoral injections in parenchymatous organs (e.g. liver, spleen, adrenal gland, pancreas) are not allowed)
  Interventions: Drug: IMP321
- Solid tumors + peritoneal carcinomatosis (Experimental): Biweekly intra-peritoneal, escalating doses of IMP321 (1 mg, 3 mg, 6 mg, 12 mg and 30 mg)
  Interventions: Drug: IMP321
- Solid tumors + chemotherapy (Experimental): Subcutaneous (s.c.) injections with the optimal dose of IMP321 defined in the AIPAC trial for a maximum of 24 weeks
  Interventions: Drug: IMP321
- NSCLC + Avelumab/IMP321 therapy (Experimental): Avelumab and IMP321 as follows:
  * 800 mg avelumab every 2 weeks i.v. (for a maximum of 24 cycles [48 weeks])
  * 6 mg (cohort 1) or 30 mg (cohort 2) IMP321 every 2 weeks s.c. (for a maximum of 12 cycles [24 weeks])
  Interventions: Drug: IMP321; Drug: Avelumab
- Urothelial carcinoma + Avelumab/IMP321 combination therapy (Experimental): Avelumab and IMP321 as follows:
  • 800 mg avelumab every 2 weeks i.v. and 30 mg IMP321 every 2 weeks s.c. for a maximum of 24 cycles [12 months]
  Interventions: Drug: IMP321; Drug: Avelumab

INTERVENTIONS:
Drug: IMP321 — LAG-3Ig fusion protein, highly potent activator of antigen presenting cells
  Other Names: LAG-3Ig fusion protein; efti; eftilagimod alfa
Drug: Avelumab — Avelumab i.v.
  Arms: NSCLC + Avelumab/IMP321 therapy; Urothelial carcinoma + Avelumab/IMP321 combination therapy

SUMMARY:
This phase I trial aims to investigate a potential enhancement of IMP321 immune-activating effects by new routes of administration: direct injection of IMP321 into the tumor tissue; intra-peritoneal therapy; combination of chemotherapy and/or immunotherapy/targeted therapy with active immunotherapy

DETAILED DESCRIPTION:
Up to now, IMP321 is solely administered by sub-cutaneous injection (e.g. on the anterior face of the thigh). In this study, we investigate whether a direct injection of IMP321 into the tumor tissue will be a useful option to improve anti-tumor immune response by placing the immune-therapeutic agent in direct vicinity of immune infiltrates in the tumor bed. This bypasses processes necessary for drug delivery to cells of solid tumors following systemic administration, like transport within vessels, transport across vasculature walls into surrounding tissues, and - in cases of peritoneal metastases - transport through the interstitial space within a tumor. For the latter case, we will also explore if an intra-peritoneal therapy represents a feasible alternative by means of delivering high drug concentrations directly to tumors located in the peritoneal cavity.

Furthermore, we will explore the possibility to extend the positive results obtained by subcutaneous injections of IMP321 in metastatic renal cell and breast carcinomas to further solid tumor entities e.g. non-small cell lung cancer (NSCLC) and urothelial carcinoma. In this part of the study, patients will be treated with the standard-of-care (SOC) chemotherapy and/or immunotherapy/targeted therapy for their tumor entity along with subcutaneous injections of IMP321.

ELIGIBILITY:
Inclusion criteria:

1. Histologically confirmed locally advanced (not manageable with curative intent) or metastatic solid tumor Specification for Stratum C: Only patients with NSCLC adenocarcinomas, (squamous or adenosquamous not permitted) who are scheduled to receive platin + pembrolizumab + pemetrexed standard treatment (only for Stratum C) Specification for Stratum E: Including only metastatic or irresectable locally advanced urothelial carcinomas - also refer to IC#14 below (only for Stratum E)
2. Tumor is accessible for repeated injections and biopsies (only for Stratum A)
3. Peritoneal carcinomatosis (only for Stratum B)
4. Patient failed standard therapy or refused standard therapy or is intolerable towards standard therapy (Strata A, B, and D) or who receives Standard-of-Care first line treatment comprising platin + pembrolizumab + pemetrexed (only for Stratum C)
5. Patient has not received more than 4 prior lines of therapy. Neoadjuvant/adjuvant treatment is not counted unless progression occurs <6 months after completion of the treatment. In these cases, neoadjuvant/adjuvant treatment is counted as one prior line (only for Stratum D).

   Specification for Stratum C: Only patients receiving first line Standard-of-Care therapy (platin + pembrolizumab + pemetrexed; only for Stratum C) Specification for Stratum E: Refer to IC#14 below with regards to previous lines of therapy; only for Stratum E) Note exclusion criterion #7 on exclusion of defined previous cancer immunotherapy (only for Strata D)
6. Patients ≥ 18 years. Patients in reproductive age must be willing to use highly effective contraception during the study and 4 months after the end of the study (appropriate contraception is defined as combined (estrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation, progestogen-only hormonal contraception associated with inhibition of ovulation, intrauterine device (IUD), intrauterine hormone-releasing system (IUS), vasectomized partner, bilateral tubal occlusion, sexual abstinence. If an oral contraception is used, a barrier method of contraception (e.g. male condom, female condom, cervical cap, diaphragm, contraceptive sponge) has to be applied additionally.). Female patients with childbearing potential need to have a negative pregnancy test within 7 days before study start.
7. ECOG 0 or 1
8. Adequate hematological, hepatic and renal function parameters:

   * ANC (absolute neutrophil count) ≥ 1,500/µL
   * Leukocytes ≥ 3,000/µL
   * Platelets ≥ 75,000/µL (for Stratum D: ≥ 100,000/µL)
   * Serum creatinine ≤ 1.5 x upper limit of normal, or GFR ≥ 50 mL/min (not applicable for patients not eligible for platinum-based therapy in Stratum E)
   * Bilirubin ≤ 1.5 - 3 x upper limit of normal (for Stratum D: ≤ 1.5 x ULN)
   * AST and ALT ≤ 3 x upper limit of normal (≤ 5 x if liver metastases are present) (for Stratum D: AST and ALT ≤ 2.5 x ULN; ≤ 5 x if liver metastases are present)
   * Alkaline phosphatase ≤ 6 x upper limit of normal
   * Hemoglobin ≥ 9 g/dL
9. Adequate coagulation functions as defined by International Normalized Ratio (INR) ≤ 1.5, and a partial thromboplastin time (PTT) ≤ 5 seconds above the ULN (unless receiving anticoagulation therapy). Patients receiving warfarin/ phenprocoumon must be switched to low molecular weight heparin (new oral anticoagulants (NOACs) are permitted) and have achieved stable coagulation profile.
10. Patient able and willing to provide written informed consent and to comply with the study protocol and with the planned surgical procedures
11. Evidence of measurable disease as defined by RECIST v1.1 (only for Strata C, D and E) or assessable disease as defined by RECIST v1.1 (only for Stratum C)
12. Expected survival > 3 months
13. Resolution of toxicity associated with prior or current therapy to grade <2 (except for alopecia and transaminases in case of liver metastases)
14. Patient is eligible if one of the following settings applies (only for Stratum E):

    * did suffer disease progression during/up to 3 months after pembrolizumab and enfortumab vedotin based first-line therapy and did receive at least 3 cycles of platinum based chemotherapy without displaying disease progression and are intended for Avelumab and Eftilagimod alpha as second-line maintenance therapy
    * did receive at least 3 cycles of platinum based chemotherapy without displaying disease progression and are intended for Avelumab and Eftilagimod alpha as first-line maintenance therapy

Exclusion criteria:

1. Inability to understand the aims of the study and/or protocol procedures
2. Bleeding ulcerative tumors or tumors requiring intratumoral injections of study drug into parenchymatous organs such as, but limited to liver, spleen or pancreas (only for Stratum A)
3. Patients with contraindication versus a laparoscopy or refusing a laparoscopy (only for Stratum B)
4. Hypersensitivity towards eftilagimod alpha, avelumab (only for Strata D and E) or any ingredient of the injection/infusion solutions
5. History of severe allergic, anaphylactic, or other hypersensitivity reactions to chimeric or humanized antibodies or fusion proteins
6. Any concurrent other antineoplastic treatment including irradiation, or targeted small molecule therapy, or biological cancer therapy. (only Strata A, Band D)
7. Prior PD-1/PD-L1 targeted therapy (only for Strata D).
8. Cirrhosis of the liver (Child > Grade A), pronounced alcohol abuse with anticipated detoxification, severe pulmonary infection with considerable reduction of pulmonary function
9. Clinically significant active coronary heart disease, cardiomyopathy or congestive heart failure, NYHA III-IV (for Stratum D: ≥ NYHA II) within 6 months prior to first dose of study treatment including: myocardial infarction, severe/unstable angina, ongoing cardiac dysrhythmias of current NCI CTCAE version Grade >2, atrial fibrillation of any grade, coronary/peripheral artery bypass graft, symptomatic congestive heart failure, cerebrovascular accident including transient ischemic attack, ventricular arrhythmias requiring medication or symptomatic pulmonary embolism
10. Cerebral or leptomeningeal metastases Note: Subjects with previously treated brain metastases may participate if they meet the following criteria: 1) are stable for at least 28 days prior to the first dose of study treatment and if all neurologic symptoms returned to baseline; 2) have no evidence of new or enlarging brain metastases; and 3) have not been using steroids for at least 7 days prior to first dose of study treatment. This exception does not include carcinomatous meningitis which is excluded regardless of clinical stability.
11. Chronic inflammatory bowel disease
12. Active infection requiring systemic therapy at the start of study treatment or chronic infection or serious intercurrent infection within 4 weeks prior to first dose of study treatment
13. QTcF >480 ms, family or personal history of long or short QT syndrome, Brugada syndrome or known history of QTc prolongation, or Torsade de Pointes (TdP)
14. Uncontrolled electrolyte disorders that can worsen the effects of a QTc-prolonging drug (e.g., hypocalcaemia, hypokalaemia, hypomagnesemia)
15. Positive test for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome. Testing is not required in the absence of history.

    Participants with known human immunodeficiency virus (HIV) infections are eligible if the following criteria are met:
    1. If clinically indicated participants must be stable on antiretroviral therapy (ART) for at least 4 weeks and agree to adhere to ART. If not clinically indicated, consult Lead Investigator.
    2. Participants with HIV infection should have no evidence of documented multidrug resistance that would prevent effective ART.
    3. Have an HIV viral load of < 400 copies/mL at Screening.
    4. If prophylactic antimicrobial drugs are indicated, patient may still be considered eligible upon agreement with the Lead Investigator
16. Active hepatitis B (defined as having a positive hepatitis B surface antigen [HBsAg] test) or hepatitis C Note: Patients with past hepatitis B virus (HBV) infection or resolved HBV infection (defined as having a negative HBsAg test and a positive antibody to hepatitis B core antigen antibody test) are eligible. Note: Patients positive for hepatitis C virus (HCV) antibody are eligible only if polymerase chain reaction testing is negative for HCV ribonucleic acid (RNA). Testing is not required in the absence of history.
17. History or evidence of interstitial lung disease, active non-infectious pneumonitis or active tuberculosis
18. Active or prior autoimmune disease requiring immunosuppressive therapy that might deteriorate when receiving an immunostimulatory agent. Patients with diabetes type I, vitiligo, psoriasis, or hypo- or hyperthyroid disease not requiring immunosuppressive treatment are eligible.
19. Known history of immune-mediated colitis, pneumonitis, pulmonary fibrosis (only for Strata D and E).
20. Administration of a live, attenuated vaccine (including Covid-19 vaccination with live, attenuated vaccine) within four weeks prior to start of treatment or anticipation that such a live attenuated vaccine will be required during the remainder of the study.
21. Any condition requiring continuous systemic treatment with either corticosteroids (>10 mg daily prednisone equivalents) or other immunosuppressive medications within 4 weeks prior to first dose of study treatment. Intranasal, inhaled or topical steroids, eye drops or local steroid injection (e.g., intra-articular injection), steroids as premedication for hypersensitivity reactions (e.g., computed tomography [CT] scan premedication) and physiological replacement doses of up to 10 mg daily prednisone equivalent are permitted in the absence of active autoimmune disease.
22. Treatment with systemic immunostimulatory agents (including but not limited to interferons or interleukin-2) within four weeks or five half-lives of the drug, whichever is shorter, prior to start of study treatment
23. Any previous venous thromboembolism > National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) Grade 3 within the last 6 months
24. Past history of severe allergic episodes and/ or Quincke's oedema
25. Prior organ transplantation or stem cell transplantation
26. On-treatment participation in another clinical study in the period 30 days prior to start of study treatment and during the study
27. Patients in a closed institution according to an authority or court decision
28. Pregnancy or lactation
29. Planned intratumoral injections in parenchymatous organs (e.g. liver, spleen, adrenal gland, pancreas)
30. Life-threatening illness unrelated to cancer
31. History of irAEs of CTCAE Grade 4 requiring steroid treatment (only for Strata C, D and E)
32. Persisting toxicity related to prior therapy (NCI CTCAE current version Grade > 1); however, alopecia, sensory neuropathy Grade ≤2, or other Grade ≤2 AEs not constituting a safety risk based on investigator's judgment are acceptable (only for Strata D and E)
33. Other severe acute or chronic medical conditions, psychiatric conditions including recent (within the past year) or active suicidal ideation or behavior; or laboratory abnormalities that may increase the risk associated with study participation or study treatment administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the patient inappropriate for entry into this study.
34. Patients with a druggable genetic alteration with an indication for targeted therapy (e.g. erdafitinib) (only for Stratum E)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2017-08-15 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Feasibility rate | 10 weeks of treatment + 2 weeks of safety observation period
  Rate of patients receiving the protocol treatment without occurrence of a dose limiting toxicity

SECONDARY OUTCOMES:
Incidence and severity of adverse events according to CTC criteria | 12 months of treatment + 12 months of Follow Up
  Incidence and severity of adverse events according to the current National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE).
Response | 12 months of Follow Up
  Objective response rate according to RECIST 1.1 and endoscopic response criteria
Progression free survival | 12 months of Follow Up
  PFS will be measured as time from inclusion until disease progression or death of any cause
Overall survival | 12 months of Follow Up
  OS will be measured as time from inclusion to death of any cause
Immune response in whole blood and tumor tissue | 12 months of treatment + 12 months of Follow Up
  Peripheral blood monocyte number and CD8 T-cell number, associated activation markers, tumor-infiltrating immune cells

CONTACTS AND LOCATIONS:
Overall Officials: Thorsten Götze, MD, Principal Investigator — Institute of Clinical Cancer Research (IKF), UCT Frankfurt, Germany
Locations (12):
- Germany (12):
  - Helios Klinikum Bad Saarow, Bad Saarow
  - Kliniken der Stadt Köln gGmbH, Studienzentrum der Lungenklinik, Krankenhaus Merheim, Cologne
  - Universitätsklinikum Essen, Essen
  - Agaplesion Markus Krankenhaus Frankfurter Diakonie Kliniken gGmbH, Frankfurt
  - Krankenhaus Nordwest, Frankfurt
  - Universität Gießen und Marburg GmbH, Giessen
  - Hämatologisch Onkologische Praxis Eppendorf (HOPE), Hamburg
  - Marienhospital Herne, Klinik der Ruhr Universität Bochum, Klinik für Urologie, Herne
  - Universitätsmedizin der Johannes Gutenberg-Universität Mainz, Mainz
  - Universitätsklinikum Tübingen, Tübingen
  - Universitätsklinikum Ulm, Early Clinical Trials Unit (ECTU), Ulm
  - Helios Dr. Horst Schmidt Klinikum Wiesbaden, Wiesbaden

IPD SHARING:
Plan to Share IPD: No
No IPD will be shared.